CLINICAL TRIAL: NCT06113055
Title: Randomised, Double Blind, Placebo-controlled Trial of L-serine in Hereditary Sensory Neuropathy Type 1.
Brief Title: Hereditary Sensory Neuropathy Serine Trial
Acronym: SENSE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1006207
Record Dates: First submitted 2023-10-12; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Hereditary Sensory Neuropathy Type I
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — Serine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-serine (Active Comparator): L-serine white or almost white crystalline powder or colourless crystal formulation which will be dissolved in water and administered orally.
  The dose will be weight based: 400mg/kg/day (total daily dose).
  Interventions: Drug: L-serine
- Dextrose (Placebo Comparator): Dextrose monohydrate powder: monohydrate form of crystalline D-glucose (dextrose) consisting of odourless, multi-granular white crystals.
  The dose will be weight based: 400mg/kg/day (total daily dose).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-serine — Active comparator
  Arms: L-serine
Drug: Placebo — Placebo comparator
  Arms: Dextrose

SUMMARY:
This is a randomised double-blind placebo-controlled trial of L-serine in Hereditary Sensory Neuropathy type 1 (HSN1) due to variants in SPTLC1/2 gene.

This is a single-centre study being conducted at the National Hospital for Neurology and Neurosurgery, London UK.

The SENSE trial will test whether L-serine is an effective drug treatment to slow or stop disease progression in HSN1 due to variants in the SPLTLC1 or SPTLC2 gene. The other aim is to assess if Magnetic Resonance Imaging (MRI) can accurately detect the changes which occur in the muscles of people who have HSN1.

DETAILED DESCRIPTION:
Hereditary Sensory Neuropathy (HSN) represents a subgroup of disorders called Charcot Marie Tooth (CMT) disease. Hereditary Sensory Neuropathy Type 1 (HSN1) is the most common subtype. It is a rare autosomal dominant (AD) neuropathy characterised by severe sensory and motor involvement for which there is no current treatment. HSN1 secondary to SPTLC1/2 mutations is the commonest type of HSN. The neuropathy is slowly progressive with onset between the second and fifth decade. The profound sensory involvement is associated with painless ulcers, recurrent osteomyelitis, and amputations. The neuropathy is very painful and pain medications are rarely fully efficacious. Motor involvement invariably follows leading to significant disability. HSN1 is due to mutations in the SPTLC1 and more rarely SPTLC2 genes which encode for the first two (out of 3) subunits of the enzyme serine palmitoyl transferase (SPT) which catalyses the first and rate limiting step in de novo sphingolipid biosynthesis. Mutations in SPTLC1 and SPTLC2 cause the neuropathy by a gain of function mechanism as mutations alter the substrate specificity of SPT whereby alanine and glycine are preferred over the canonical serine resulting in the production of neurotoxic deoxysphingolipids (DSBs).

This single-site double-blinded placebo-controlled trial will investigate whether L-serine is efficacious in the treatment of HSN1 due to SPTLC1/2 mutations.

The primary objective is to identify if treatment with L-serine is efficacious in the treatment of HSN1 due to SPTLC1/2 mutations compared to treatment with placebo. A major objective will be to validate the use of the MRC Muscle Fat Fraction protocol as a primary outcome measure in inherited neuropathies trials. The MRC Muscle Fat Fraction protocol has been shown to be a responsive biomarker in natural history studies in several inherited neuropathies including HSN, but not previously in clinical trials. Regardless of the efficacy outcome, the trial will assess the feasibility of MRI as an outcome measure in a clinical trial setting, and comparison of the results in the placebo arm to previous natural history study data will validate the translation of natural history results to the clinical trial setting.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥ 18 with genetically proven HSN1 due to SPTLC1/2 mutations.
* Participants must be able to undergo an MRI scan without sedation.
* Participants must be able to complete the Charcot Marie Tooth Neuropathy Score (CMTNS)
* Participants must have a CMTES ≤ 26
* Female participants of childbearing potential must agree to use a highly effective method of contraception from the time consent is signed until six days after treatment discontinuation (this is to allow for medication wash out post treatment discontinuation).
* Participants must be willing and able to provide written informed consent.

Exclusion Criteria:

* Participants have undergone foot surgery in the 6 months prior to trial enrolment or are due to undergo foot surgery during the trial
* Participants have a history of nephrolithiasis
* Participants have another medical condition which precludes them from having an MRI scan or from completing the CMTNSv2
* Participants with known diagnosis of another neuromuscular disease
* Participants with diabetes
* Females who are planning pregnancy or are pregnant or breastfeeding.
* Patient taking regular L-serine supplementation within 6 months of study commencement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
MRC Muscle Fat Fraction protocol | 12 months
  The primary outcome measure will be the mean difference in change from baseline lower limb muscle fat fraction at the severity appropriate anatomical level measured by MRI over 12 months between L-serine treated and placebo treated groups. The primary outcome has units of percentage fat fraction (%FF) and is a continuous variable.

SECONDARY OUTCOMES:
Secondary outcome measures | 12 months
  Charcot Marie Tooth Neuropathy Score (CMTNS) v2 and v2-Rasch
Secondary/Exploratory outcome measures | 12 months
  plasma neurofilament light chain levels
Secondary/Exploratory outcome measures | 12 months
  plasma deoxysphingolipid levels
Secondary/Exploratory outcome measures | 12 months
  thigh intraepidermal nerve fibre density
Secondary outcome measures | 12 months
  Charcot Marie Tooth Health Index Quality of Life Score
Secondary outcome measure | 12 months
  Neuropathic Pain Diagnostic Questionnaire
Secondary outcome measure | 12 months
  Neuropathic Pain Symptom Inventory
Secondary outcome measure | 12 months
  Brief Pain Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No